CLINICAL TRIAL: NCT01591525
Title: Diabetes Mellitus Community Based Screening in Minority Populations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ethnicity and Disease Community Empowerment Center (Other)
Collaborators: Steward Carney Hospital (Unknown); Boston Public Housing Authority (Unknown)
Responsible Party: Sponsor
Other Study IDs: EADCEC-001
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Type II Diabetes; Diabetes Mellitus
Keywords: Type II Diabetes; Minorities; Diabetes Mellitus; Community based screening
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Early Intervention, Educational

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Uncontrolled Diabetic: Individuals who were previously diagnosed with Type II Diabetes, but have a HgA1C greater than 7.0%
  Interventions: Behavioral: Education on risk factors for Type II Diabetes; Behavioral: Education on Type II Diabetes; Behavioral: Education on regular visits to a Primary Care Provider
- Newly diagnosed Type II Diabetic: Individuals who have never been diagnosed with Type II Diabetes, but have an HgA1c greater than 7.0%
  Interventions: Behavioral: Education on risk factors for Type II Diabetes; Behavioral: Education on Type II Diabetes; Behavioral: Education on regular visits to a Primary Care Provider
- Newly diagnosised pre-diabetics: Individuals who have never been diagnosed with Type II Diabetes, but have a HgA1C of 6.0%-6.9%
  Interventions: Behavioral: Education on risk factors for Type II Diabetes; Behavioral: Education on Type II Diabetes; Behavioral: Education on regular visits to a Primary Care Provider
- Controlled: Diabetic or non-diabetic individuals with RPCG of less than 130 mg/dl.
  Interventions: Behavioral: Education on risk factors for Type II Diabetes; Behavioral: Education on regular visits to a Primary Care Provider

INTERVENTIONS:
Behavioral: Education on risk factors for Type II Diabetes — one-on-one education provided by a nurse practitioner or physician
  Other Names: educational intervention
Behavioral: Education on Type II Diabetes — one-on-one education about having Type II Diabetes, the possible complications and treatment options provided by a physician.
  Other Names: educational intervention
  Groups: Newly diagnosed Type II Diabetic; Newly diagnosised pre-diabetics; Uncontrolled Diabetic
Behavioral: Education on regular visits to a Primary Care Provider — one-on-one education about the importance of visiting a primary care provider (PCP) on a regular basis. Patients are also provided a list of PCP's accepting new patients within a 3 mile radius.
  Other Names: educational intervention

SUMMARY:
The purpose of the type II diabetes (T2D) screening study is to improve diabetes care in minority communities by identifying undiagnosed and uncontrolled T2D patients, as well as help patients without a regular primary care physician (PCP) find one within their community. These goals will be achieved first through a glucose measurement. Individuals with a high glucose measurement will be confirmed with a rapid hemoglobin A1c (HgA1c) test. The HgA1c test will tell us about the patients average blood sugar over the past 3 months, which will allow us to immediately diagnose new and uncontrolled type II diabetics. All participants will fill out a survey on healthcare seeking behaviors before glucose testing. All patients who enter the study will receive education on T2D and the value of regularly visiting their PCP, and will be provided a list of PCP currently accepting new patients within a 3 mile radius. Follow-up visits at 4 and 8 months will help us determine the success this community based screening.

The investigators hypothesis is that community based screening designed with adequate education and follow-up, and performed by qualified medical professionals will improve diabetes care in minority communities as assessed through hemoglobin A1c levels over 8 months, and in the change in the number patients who visit/obtain their PCP within the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and older

Exclusion Criteria:

* Type I Diabetes.
* Women who are currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents in Boston Public Housing
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Lamb, MA, Study Director — Ethnicity and Diseasse Community Empowerment Center; Jean Bonnet, MD, Principal Investigator — Ethnicity and Disease Community Empowerment Center; James Morgan, MD, Principal Investigator — Steward Carney Hospital
Locations (1):
- Lower Mills, Dorchester, Massachusetts, United States